CLINICAL TRIAL: NCT02428296
Title: Nonrandomized Open Label Pilot Study of Sirolimus Therapy for Segmental Overgrowth Caused by Somatic PI3K Activation
Brief Title: Study of Sirolimus Therapy for Segmental Overgrowth Caused by Somatic PI3K Activation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150120; 15-HG-0120 (Other: National Institutes of Health)
Record Dates: First submitted 2015-04-23; First posted 2015-04-28 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2018-02-14

CONDITIONS: PIK3CA-Related Overgrowth Spectrum (PROS); Growth Disorder; Genetics
Keywords: Clinical Trial; Congenital Malformations; Overgrowth; Pilot Drug Treatment Trial
MeSH Terms: conditions — Growth Disorders; Congenital Abnormalities | interventions — Sirolimus

ARMS (1):
- Patients with PIK3CA gene mutation treated with Sirolimus (Experimental): This is a single-arm, non-randomized, open-label study for the treatment of segmental overgrowth disorders (somatic PIK3CA gene mutation) with Sirolimus in thirty-nine patients.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Low dose sirolimus will be given in daily dosing to achieve trough levels of 2-6 ng/ ml.

SUMMARY:
Background:

- PIK3CA-related overgrowth spectrum (PROS) is caused by changes in the PIK3CA gene. This gene makes a protein that communicates with other proteins in the body to cause cells to grow. Alterations in PIK3CA change the chemical signals in the body and cause overgrowth in fatty, vascular and other tissues. Sirolimus is a drug that reduces the signals sent by one of the proteins in this chemical signaling pathway. Researchers want to learn whether the drug sirolimus can reduce or stabilize some of the overgrowth that patients with PROS experience.

Objectives:

- To measure how the overgrowth of patients with PROS changes over time and whether taking a drug called sirolimus can reduce or stabilize a person s overgrowth.

Eligibility:

- People ages 3 to 65 years old with a confirmed mutation or alteration of the PIK3CA gene in the person s affected tissues (a somatic mutation).

Design:

* Participants will be screened with medical history and genetic counseling.
* First 6 months: Participants will have their overgrowth monitored.
* Next 6 months: Participants will take sirolimus once or twice a day.
* Participants will have to visit the clinic several times, and stay in the area for 4 to 5 days each time.
* Participants will have a one month-long visit to the clinic.
* During clinic visits, participants will have:
* Blood and urine tests.
* Photographs of their physical features.
* Scans, including an MRI and DEXA, and possibly x-rays and CT scans.
* For the MRI and CT scans, participants will lie in a machine that takes pictures of their body.
* The DEXA involves a small amount of radiation.
* They may have:
* Non-invasive heart function tests.
* Lung function tests.
* Participants will have several blood and urine tests between visits.
* Participants will complete surveys and keep a diary of their treatment and side effects.
* Participants may visit other health specialists or undergo other tests based on side effects.
* One month after stopping the study drug, participants will have 1 clinic visit.

DETAILED DESCRIPTION:
The primary study objective is to determine the likely size of sirolimus treatment effect. The patient population will include male and female subjects, aged greater than or equal to 3 years and less than or equal to 65 years of age with segmental overgrowth identified to have clinical and molecular findings of somatic PIK3CA gene mutation. The planned study size will be ten patients seen at the NIHCC. An additional 20 patients will be contributed by two other centers, who will be responsible for the conduct of the proposed research at their site, but the study procedures and dosing schedule will be identical to enable pooling of results for statistical analyses. The study design will be a nonrandomized, open label, phase II pilot study of sirolimus treatment. As patients have highly variable clinical presentations, and there are no established evidence-based methodologies for measuring serial changes in growth, the aim of this pilot study is to establish the optimal methodology for evaluating changes in growth to inform the design of a future randomized controlled trial, in addition to determining treatment effect size, and evaluating safety and toxicity of low dose sirolimus. Overall desired outcome will be reduced size of affected body part, and measures will include: reduction in affected tissue (fibroadipose or bone) size by clinical exam measurement and by radiological studies (MRI area measurements and/or DXA study measurements of fat).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age: greater than or equal to 3 years to less than or equal to 65 years
* Male or Female
* Confirmed PIK3CA somatic mutation
* Measurably progressive overgrowth, in current progression or with clinical history of overgrowth progression
* Adequate Bone Marrow Function Defined as:

  * Peripheral absolute neutrophil count (ANC) greater than or equal to 1500/microliter, except for those participants with an absolute neutrophil count (ANC) of 1000-1500, caused by a benign condition associated with moderately decreased neutrophils known as Benign Ethnic Neutropenia (BEN), d those who have an ANC of 1000-1500 caused by a confirmed infection, which resolves with treatment of infection to greater than or equal to 1500.
  * Platelet count less than or equal to 100,000/microliter
  * Hemoglobin less than or equal to 10.0 gm/dL
* Adequate Renal Function Defined as:
* A serum creatinine based on age as follows:

  * Age (years) [Maximum Serum Creatinine (mg/dl)]
  * Less than or equal to 5 [0.8 mg/dl]
  * 5 less than age less than or equal to10 [1.0 mg/dl]
  * 10 less than age less than or equal to 15 [1.2 mg/dl]
  * Less than 15 [1.5 mg/dl]
* OR a creatinine clearance or radioisotope GFR greater than or equal to 70ml/min/1.73 m2

  * Adequate Liver Function Defined As:

    * Bilirubin (sum of conjugated + unconjugated) less than or equal to 1.5 x upper limit of normal (ULN) for age, and
    * SGPT (ALT) less than or equal to 5 x upper limit of normal (ULN) for age, and
    * Serum albumin greater than or equal to 2 g/dL.
  * Fasting LDL Cholesterol:

    * Patients must have a fasting LDL cholesterol of less than or equal to 160 mg/d
    * All women of childbearing potential and all sexually active male patients must agree to use effective contraception
    * Adolescent (15-17 year old) participants who are fluent in English and can thereby complete the pediatric self-report questionnaires and communicate well with the study team but whose parent(s) and/or legal guardian are primarily Spanish-speaking.

EXCLUSION CRITERIA:

The participant may not enter the study if ANY of the following apply:

* Age less than 3 years or greater than 65 years
* Pregnant or breastfeeding
* Women and men of reproductive age without an effective method of contraception (during treatment and up to 12 weeks after sirolimus discontinuation)
* Hypersensitivity to sirolimus or any of the excipients
* Any current medical disorder or medication likely to impair ability to follow the study protocol safely and effectively
* Incapacity to give informed consent
* Sirolimus treatment in the prior 4 weeks
* If less than 3 months post-surgery
* Prior malignancy or ongoing investigations for malignancy
* Active skin infections requiring antibiotics or anti-viral medication
* HCV/HBV/HIV seropositivity
* Previous/ active MTB infection
* Pneumonitis
* Research radiation exposure within previous 12 months
* Adult participants or participants under the age of 15 years with insufficient English language proficiency to complete informed consent and quality of life measures

We propose to restrict participation in this study to those with sufficient English language skills to complete the quality of life measures we will employ among all three study sites, as many of the specific quality of life measures we are employing at the NIH only are not available in other languages.

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-04-23; Primary Completion 2018-02-14 (Actual); Study Completion 2018-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim M Keppler-Noreuil, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Lindhurst MJ, Parker VE, Payne F, Sapp JC, Rudge S, Harris J, Witkowski AM, Zhang Q, Groeneveld MP, Scott CE, Daly A, Huson SM, Tosi LL, Cunningham ML, Darling TN, Geer J, Gucev Z, Sutton VR, Tziotzios C, Dixon AK, Helliwell T, O'Rahilly S, Savage DB, Wakelam MJ, Barroso I, Biesecker LG, Semple RK. Mosaic overgrowth with fibroadipose hyperplasia is caused by somatic activating mutations in PIK3CA. Nat Genet. 2012 Jun 24;44(8):928-33. doi: 10.1038/ng.2332. PMID 22729222
- [Background] Keppler-Noreuil KM, Rios JJ, Parker VE, Semple RK, Lindhurst MJ, Sapp JC, Alomari A, Ezaki M, Dobyns W, Biesecker LG. PIK3CA-related overgrowth spectrum (PROS): diagnostic and testing eligibility criteria, differential diagnosis, and evaluation. Am J Med Genet A. 2015 Feb;167A(2):287-95. doi: 10.1002/ajmg.a.36836. Epub 2014 Dec 31. PMID 25557259
- [Background] Keppler-Noreuil KM, Sapp JC, Lindhurst MJ, Parker VE, Blumhorst C, Darling T, Tosi LL, Huson SM, Whitehouse RW, Jakkula E, Grant I, Balasubramanian M, Chandler KE, Fraser JL, Gucev Z, Crow YJ, Brennan LM, Clark R, Sellars EA, Pena LD, Krishnamurty V, Shuen A, Braverman N, Cunningham ML, Sutton VR, Tasic V, Graham JM Jr, Geer J Jr, Henderson A, Semple RK, Biesecker LG. Clinical delineation and natural history of the PIK3CA-related overgrowth spectrum. Am J Med Genet A. 2014 Jul;164A(7):1713-33. doi: 10.1002/ajmg.a.36552. Epub 2014 Apr 29. PMID 24782230
- [Result] Parker VER, Keppler-Noreuil KM, Faivre L, Luu M, Oden NL, De Silva L, Sapp JC, Andrews K, Bardou M, Chen KY, Darling TN, Gautier E, Goldspiel BR, Hadj-Rabia S, Harris J, Kounidas G, Kumar P, Lindhurst MJ, Loffroy R, Martin L, Phan A, Rother KI, Widemann BC, Wolters PL, Coubes C, Pinson L, Willems M, Vincent-Delorme C; PROMISE Working Group; Vabres P, Semple RK, Biesecker LG. Safety and efficacy of low-dose sirolimus in the PIK3CA-related overgrowth spectrum. Genet Med. 2019 May;21(5):1189-1198. doi: 10.1038/s41436-018-0297-9. Epub 2018 Oct 1. PMID 30270358
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-HG-0120.html

RESULTS

PARTICIPANT FLOW:
Groups:
- PIK3CA-Related Overgrowth Spectrum Patients: Participants were assessed for sirolimus efficacy at week 0 (before the run-in phase), week 26 (after the run-in phase and before treatment), and at week 52 (after 26 weeks of treatment).
  Pharmacokinetic data for sirolimus for children and adults with renal transplants informed dosing algorithms. A target sirolimus plasma concentration of 2-6ng/ml was selected based on in vitro preclinical studies off-label clinical experience, and with the aim of minimizing AEs.
Period: Overall Study
Arm/Group | PIK3CA-Related Overgrowth Spectrum Patients
Started | 39
Treated | 39
Completed | 30 (Number of participants who completed the full course of treatment.)
Not Completed | 9
Not completed — Adverse Event | 7
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | PIK3CA-Related Overgrowth Spectrum Patients
Number analyzed (Participants) | 39
Age, Continuous [Mean (Full Range); unit: years] | 16.6 [3 to 48]
Age, Customized [Count of Participants; unit: Participants]
  Age: 3-16 years | 23
  Age: 17-48 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13
  France | 15
  United Kingdom | 11

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Unaffected and Affected Fibrofatty Tissue Measured by DXA
Description: The primary outcome measures will use quantitative DXA scan of the affected and unaffected body part (s) to demonstrate negative change in fibrofatty, muscular, and/or bony overgrowth.
  Absolute volumes of affected and unaffected tissue at week 0 (designated X), week 26 (designated Y), and week 52 (designated Z), were compared by taking the difference between the mean value obtained during the run-in period and the mean value obtained during the treatment period. Tissue volume changes (week 0-26 and week 26-52) were designated "DELTA," and the percent change "% Change." Percent change for the untreated period was [100(Y-X/X)], and for the treated period [100(Z-Y/Y)].
Time Frame: Run-in (0-26 weeks), treatment (26-52 weeks)
Population: The anatomy of 23 patients permitted DXA analysis of affected versus unaffected tissue.
Measure: Mean (Standard Deviation); unit: mean percentage change in tissue volume
Groups:
- Affected Tissue: Affected sites were defined by clinical observation.
- Unaffected Tissue: Unaffected sites showed no overgrowth, nor evidence of skin or vascular abnormalities.
Arm/Group | Affected Tissue | Unaffected Tissue
Number analyzed (Participants) | 23 | 23
mean percentage change in tissue volume
  Run-in period | 7.9 (12.8) | 4.8 (9.7)
  Treatment period | 0.71 (10.2) | 6.5 (12.3)
  Change in mean percentage change of tissue volume | -7.2 (16.0) | 1.7 (11.5)

2. Primary Outcome: Percent Change in Unaffected and Affected Fibrofatty Tissue Measured by MRI Scan
Description: The outcome was measured as a percent change in tissue volume between the treatment period and run-in period.
  For volume calculation, IDEAL fat (Dixon sequence) images were visualized using volumetric software (SliceOmatic, TomoVision, Magog, Canada). Morphology segmentation was performed through computation of watershed gradients. Tissues (fat, muscle, bone, and blood vessel) were manually defined and software was used to generate a surrogate of tissue volume using five slices, with manual adjustments where required.
  Absolute volumes of affected and unaffected tissue at week 0 (designated X), week 26 (designated Y), and week 52 (designated Z), were compared. Tissue volume changes (week 0-26 and week 26-52) were designated "DELTA," and the percent change "% Change." Percent change for the untreated period was [100(Y-X/X)], and for the treated period [100(Z-Y/Y)].
Time Frame: Run-in (0-26 weeks), treatment (26-52 weeks)
Population: Ten MRI series were analyzed. Only six of ten MRI series that were eligible for analysis included both affected and unaffected sites (the remaining only measured affected tissue).
Measure: Mean (Standard Deviation); unit: percentage of tissue volume change
Arm/Group | Affected Tissue | Unaffected Tissue
Number analyzed (Participants) | 10 | 6
percentage of tissue volume change | -3.7 (12.3) | 0 (16.7)

3. Secondary Outcome: Mean Sirolimus Doses to Achieve the Target Plasma Concentration
Description: To establish optimal sirolimus dosing algorithms for a future RCT.
Time Frame: Between 6 months and 12 months
Population: All patients were analyzed to determine at which dose the patient would reach the target plasma concentration.
Measure: Mean (95% Confidence Interval); unit: mg/day
Arm/Group | PIK3CA-Related Overgrowth Spectrum Patients
Number analyzed (Participants) | 39
mg/day
  Adults: number analyzed (Participants) | 17
  Adults | 1.2 [1.1 to 1.3]
  Children: number analyzed (Participants) | 22
  Children | 1.16 [1.0 to 1.3]

4. Secondary Outcome: Additional Measure of Efficacy: Quality of Life Assessment
Description: The World Health Organization Quality of Life-BREF (WHOQOL-BREF) assessment measures four domains related to quality of life (physical health, psychological, social relationships, and environment) and produces both individual domain scores (0-100) a total score on a 0-100 scale (high scores indicate a better quality of life). This measure was used to assess quality of life of parents on behalf of their children, and adult subjects.
  The Pediatric Quality of Life (PedsQL) assessment is scored on a 0-100 scale (high scores indicate a better health related quality of life). This measure was used to assess quality of life of children.
  The outcomes are reported as a change in quality of life based on the change in scores from these assessments between baseline (time 0 months) and end of treatment (time 12 months).
Time Frame: baseline (0 months) and end of treatment (12 months)
Population: Children (N=15) and parents of children (N=19) were administered quality of life questionnaires. Adult subjects (N=9) were also administered quality of life questionnaires, but the scores were reported as individual domain mean scores; health total mean scores were not reported. Total score data for adults was not analyzed or reported.
Measure: Mean (95% Confidence Interval); unit: mean change in quality of life score
Arm/Group | Patients With PIK3CA Gene Mutation Treated With Sirolimus
Number analyzed (Participants) | 43
mean change in quality of life score
  Children (total health): number analyzed (Participants) | 15
  Children (total health) | -1.7 [-5.0 to 8.8]
  Parents (total health): number analyzed (Participants) | 19
  Parents (total health) | 4.9 [-0.7 to 10.4]
  Adults (physical health): number analyzed (Participants) | 9
  Adults (physical health) | 0.25 [-8.9 to 9.4]
  Adults (psychological health): number analyzed (Participants) | 9
  Adults (psychological health) | -1.25 [-7.3 to 4.8]
  Adults (social relationships): number analyzed (Participants) | 9
  Adults (social relationships) | 6.3 [-1.8 to 14.3]
  Adults (environment): number analyzed (Participants) | 9
  Adults (environment) | -7.3 [-32.5 to 17.7]

5. Secondary Outcome: Number of Hospitalizations and Surgical Interventions
Description: Tracked number of hospitalizations and surgical interventions occurring over the course of the run-in and treatment period.
Time Frame: Run-in (0-26 weeks) and treatment (27-52 weeks)
Measure: Number; unit: number of events
Arm/Group | PIK3CA-Related Overgrowth Spectrum Patients
Number analyzed (Participants) | 39
number of events
  Run-in period : Hospitalizations | 5
  Run-in period : Surgical interventions | 2
  Treatment period : Hospitalizations | 9
  Treatment period : Surgical interventions | 0

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse event definitions are consistent with the clinicaltrials.gov definitions. AEs were identified by laboratory testing, clinical examination, or self-report. Severity was graded with the CTCAE (version 4.0). All AEs and SAEs possibly, probably, or definitely related to sirolimus were reviewed by an international committee.
Arm/Group | PIK3CA-Related Overgrowth Spectrum Patients
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 12/39
Other Adverse Events (participants affected / at risk) | 31/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PIK3CA-Related Overgrowth Spectrum Patients (N=39)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Neutropenic fever (Blood and lymphatic system disorders) | 1 (1)
Constipation aggravated (Gastrointestinal disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (6)
Epstein Barr Virus (Infections and infestations) | 1 (1)
Pelvic infection (Infections and infestations) | 1 (1)
Viral meningitis (Infections and infestations) | 1 (1)
Over-medication (Injury, poisoning and procedural complications) | 1 (1)
Sirolimus hypersensitivity syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Hemarthrosis (Vascular disorders) | 1 (1)
Pulmonary embolus (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PIK3CA-Related Overgrowth Spectrum Patients (N=39)
Blood and lymphatic disorders (Blood and lymphatic system disorders) | 8 (8)
Gastrointestinal disorders (Gastrointestinal disorders) | 2 (2)
Infections and infestations (Infections and infestations) | 16 (21)
Injury, poisoning, and procedural complications (Injury, poisoning and procedural complications) | 1 (1)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 3 (3)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 (1)
Nervous system disorders (Nervous system disorders) | 2 (2)
Renal and urinary disorders (Renal and urinary disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Skin and subcutaneous disorders (Skin and subcutaneous tissue disorders) | 2 (2)
Vascular disorders (Vascular disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
Phenotypic heterogeneity; post hoc subanalyses and QoL assessments had small sample sizes; overestimation of AEs; interruption of treatment due to intercurrent AEs; asymmetric overgrowth not included in primary outcome analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/96/NCT02428296/Prot_SAP_000.pdf